CLINICAL TRIAL: NCT07293494
Title: Neurobehavioral Changes Following Spaceflight Stressors
Acronym: NeuroSTAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); University of Florida (Other); Cornell University/Weill Cornell Medical Center (Unknown); National Aeronautics and Space Administration (NASA) (U.S. Federal Agency); University of Nevada, Las Vegas (Other); Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 858402; 80JSC024NA001-NSCOR (Other Grant/Funding Number: NASA)
Record Dates: First submitted 2025-12-05; First posted 2025-12-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Stressor, Individual; Alcohol Impairment; Sleep Deprivation; Impairment, Cognitive
MeSH Terms: conditions — Stress, Psychological; Sleep Deprivation; Cognitive Dysfunction | interventions — Ethanol; Wakefulness

STUDY DESIGN:
Intervention Model Description: After an adaptation night, subjects will be exposed to the following three scenarios in various orders across the following four nights:
  1. Control night (CTRL), without any intervention;
  2. Alcohol administration (ALC), where subjects will be dosed to approximately 0.08% BAC and monitored as their BAC descends to near 0.0% before sleep;
  3. Acute total sleep deprivation (SD1&2), where subjects will remain awake for 27 hours (SD1) until a daytime 3-hour nap opportunity, followed by a recovery night sleep opportunity of 9 hours (SD2).
  Each of these three conditions occurs in a randomized and balanced fashion across the study. There are six different possible orders that a subject can be assigned to. All subjects in one group will receive the same condition at the same time.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group A: CTRL - ALC - SD1&2 (Experimental): Group A will experience the interventions in the following order, following an adaptation night sleep from 11 PM to 8 AM: Control (CTRL); Alcohol Administration (ALC); Sleep Deprivation for 27 hours (SD1) with Sleep Recovery (SD2).
  Interventions: Other: Alcohol Administration; Behavioral: Sleep Deprivation; Other: Control
- Group B: ALC - CTRL - SD1&2 (Experimental): Group B will experience the interventions in the following order, following an adaptation night sleep from 11 PM to 8 AM: Alcohol Administration (ALC); Control (CTRL); Sleep Deprivation for 27 hours (SD1) with Sleep Recovery (SD2).
  Interventions: Other: Alcohol Administration; Behavioral: Sleep Deprivation; Other: Control
- Group C: SD1&2 - CTRL - ALC (Experimental): Group C will experience the interventions in the following order, following an adaptation night sleep from 11 PM to 8 AM: Sleep Deprivation for 27 hours (SD1) with Sleep Recovery (SD2); Alcohol Administration (ALC); Control (CTRL).
  Interventions: Other: Alcohol Administration; Behavioral: Sleep Deprivation; Other: Control
- Group D: CTRL - SD1&2 - ALC (Experimental): Group D will experience the interventions in the following order, following an adaptation night sleep from 11 PM to 8 AM: Control (CTRL); Sleep Deprivation for 27 hours (SD1) with Sleep Recovery (SD2); Alcohol Administration (ALC).
  Interventions: Other: Alcohol Administration; Behavioral: Sleep Deprivation; Other: Control
- Group E: ALC - SD1&2 - CTRL (Experimental): Group E will experience the interventions in the following order, following an adaptation night sleep from 11 PM to 8 AM: Alcohol Administration (ALC); Sleep Deprivation for 27 hours (SD1) with Sleep Recovery (SD2); Control (CTRL).
  Interventions: Other: Alcohol Administration; Behavioral: Sleep Deprivation; Other: Control
- Group F: SD1&2 - ALC - CTRL (Experimental): Group F will experience the interventions in the following order, following an adaptation night sleep from 11 PM to 8 AM: Sleep Deprivation for 27 hours (SD1) with Sleep Recovery (SD2); Alcohol Administration (ALC); Control (CTRL).
  Interventions: Other: Alcohol Administration; Behavioral: Sleep Deprivation; Other: Control

INTERVENTIONS:
Other: Alcohol Administration — For the alcohol administration condition (ALC), subjects will consume alcohol within a window of approximately fifteen minutes in the morning in order to induce a blood alcohol content (BAC) level of 0.08%, in the form of 80-proof vodka mixed with fruit juice or clear, noncaffeinated soda at a 1:3 ratio. The specific dosage is determined by the Widmark formula, factoring in each individual's body weight and sex. BAC will be measured by a NHTSA-approved evidential breath testing (EBT) device, which measures breath alcohol content (BrAC, in grams per 210 liters of breath) and converts it to BAC (in g/100ml or g/dl). BAC will be measured before and after every task until subjects go to bed at 11 PM, at which point their BAC is expected to be at or close to 0.00%. Subjects will undergo an MRI (shortly after alcohol consumption at what is anticipated to be their highest level of intoxication to capture the impairing effects) and two blood draws (in the morning and afternoon).
  Other Names: Alcohol; Intoxication
Behavioral: Sleep Deprivation — For the sleep deprivation condition (SD1&2), subjects will remain awake for 27 hours from 8 AM until 11 AM the following morning (SD1). They will perform testing at regular intervals throughout the day and overnight, and they have two blood draws during the extended wake period. Subjects will undergo an MRI after approximately 25 hours of wakefulness, followed by a three-hour nap opportunity from 11 AM until 2 PM. They will then remain awake from 2 PM until 11 PM for testing and meals before returning to the standard sleep period of 11 PM to 8 AM (SD2). Caffeine will not be available to subjects during this period nor will it be available at any other time during the study.
  Other Names: Sleep Restriction; Wakefulness
Other: Control — During the control condition (CTRL), subjects will have no stressor intervention. They will not consume alcohol and they will sleep during the standard period of 11 PM to 8 AM. They will perform testing at regular intervals throughout the day. They will undergo an MRI in the morning, and have two blood draws (in the morning and afternoon).

SUMMARY:
This study aims to investigate the impairing effects of known central nervous system (CNS) stressors in a controlled environment in order to predict and mitigate analogous risks in spaceflight. Up to 56 healthy individuals aged 25-60 will spend approx. 110 hours in a laboratory, where they will be exposed to 27 hours of sleep deprivation and will consume alcohol to reach a BAC of 0.08 on a separate day. They will perform cognitive and sensorimotor tasks and undergo MRIs and blood draws.

DETAILED DESCRIPTION:
This study aims to investigate the impairing effects of known central nervous system (CNS) stressors in a controlled environment in order to predict and mitigate analogous risks in spaceflight. Up to 56 healthy individuals aged 25-60 will spend six days and five nights (24 hours a day) in a laboratory, where they will be exposed to 27 hours of sleep deprivation and will consume alcohol to reach a BAC of 0.08 on a separate day. They will also have an adaptation night, a control condition with no daytime or nighttime interventions, and a recovery night following the sleep deprivation condition. All subjects in a group will receive the three conditions (sleep deprivation, alcohol administration and control) in the same order, but this order will vary between study runs.

Subjects will perform cognitive tests and sensorimotor tasks throughout the waking periods. They will undergo one MRI and two blood draws for each of the three conditions, for a total of three MRIs and six blood draws per subject. The scans and blood draws are timed to occur near the highest predicted level of impairment in order to capture the dose-response relationship between the stressor and performance. Combined with research from parallel rodent studies performed at a partner institution where rodents are exposed to alcohol administration, sleep deprivation and radiation, these data may allow us to estimate the performance decrements associated with exposure to radiation in humans to assess the radiation risks of spaceflight.

ELIGIBILITY:
Inclusion Criteria:

* Age between 25-60 years.
* Free of psychological, psychiatric or physical conditions that preclude participation.
* BMI between 18.5 and 35.
* Self-reported regular sleep schedule; able to maintain their sleep schedule during the course of the study.
* Self-reported sleep duration of 6-8.5 h per night (verified by daily logs).
* Ability to read/write English.
* Able to stand unassisted for up to 10 minutes at a time and able to lift arms above head.

Exclusion Criteria:

* Alcohol or drug abuse in the past year based upon history and urine toxicology screen.
* Potential alcohol abuse or heavy drinking in the past year, based on self-report (AUDIT-C Q2 score above 1 or Q3 score above 2).
* Alcohol-naive based on self-report (AUDIT-C Q1 score of 0).
* Allergies, conditions or circumstances that preclude alcohol consumption, including use of medication or supplements (prescription or over the counter) that could interfere with study participation or make it hazardous for a subject to partake (e.g., anticholinergics; antipsychotics; lithium; psychotropic drugs not otherwise specified), or for which alcohol consumption should be limited or avoided (e.g. items identified on NIAAA's 'Harmful Interactions' list).
* Cultural or personal beliefs that preclude alcohol consumption.
* Body Mass Index ≤18.5 or ≥ 35.
* Current smoker/tobacco user or using nicotine replacement therapy. Those that have been nicotine-free for ≥ 30 days may be included.
* Excessive caffeine consumption (> 650mg/day combining all caffeinated drinks regularly consumed during the day).
* Acute, chronic, or debilitating medical conditions, major Axis I psychiatric illness based on history, physical exam, blood and urine chemistries; or self-reported history of neurological, psychiatric, or other medical condition that precludes participation, such as nervous system disorders, dementia, chronic migraines, or epilepsy; panic, bipolar or schizoaffective disorder; sleep disorders including insomnia, narcolepsy and obstructive sleep apnea; liver, kidney or heart disease, hypertension; infectious diseases; diabetes; or any other conditions for which medical monitoring is advised and which may require medications and/or lifestyles that preclude alcohol consumption and/or sleep disruption.
* Current depression as determined on the Beck Depression Inventory (Beck, 1996), by either a total score of 19 or higher or a response greater than 0 on Q9 (suicidality).
* Cardiovascular, gastrointestinal, or musculoskeletal problems, or other major conditions such as organ failure, cancer or patients requiring oxygen.
* Prior history or diagnosis of any sleep disorder including Obstructive Sleep Apnea (AHI ≥15 events/hour) - from ambulatory or in lab polysomnography; Restless legs syndrome or periodic limb movement disorder; Insomnia; Parasomnia; High Risk of OSA based on STOP-BANG Questionnaire ("yes" on at least 4 of 8 questions); High Risk of Restless Legs Syndrome (RLS) based on Cambridge-Hopkins Screening questionnaire; High Risk of Insomnia based on Insomnia Severity Index (score of 22 or higher).
* Current use or use within the past month of a prescription or over-the-counter sleep medication or stimulant (based on self-report or review with a study clinician).
* History of potential MRI contraindications, including: tinnitus; sensorineural hearing loss > 30 dB; pace maker or internal defibrillator; metallic implants (e.g. orthopedic plates after bone fractures, joint replacements, surgical staples or clips, artificial heart valves, stents, cava filters); metallic splinters (e.g. after an accident or due to war injury); non-removable dental brace; Tattoo (some tattoo inks contain metallic particles); permanent make-up; non-MRI compatible intrauterine contraceptive device; cochlear implant (implanted hearing device); medication pump; acupuncture needle; other foreign bodies/objects which are non-removable; pregnancy (or its possibility); previous brain and/or heart surgery.
* History of severe motion sickness, based on self-report or driving simulator response.
* Pregnant or currently breast feeding. People that menstruate will have a pregnancy test performed via urine sample during screening, as those that are currently pregnant are unable to participate in the study.
* Individuals who self-report severe contact dermatitis or allergy to bandages, silicone, nickel or silver.
* Currently working night, swing, split or rotating shift.
* Planned travel across more than one time zone within 7 days of the scheduled study start date.
* Habitual daytime napping.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Psychomotor Vigilance Task (PVT) lapses | From Study Day 2 through Study Day 6 (to include each of the three conditions: ALC, CTRL, SD1&2).
  The number of lapses in the Psychomotor Vigilance Task (PVT) in the Cognition battery, a 3-minute task that records reaction times to visual stimuli and has been validated as a sensitive measure of vigilant attention. Subjects are instructed to monitor a blank box on the screen, and to hit the space bar once a millisecond counter appears in the box and starts incrementing. The box displays the reaction time for one second then resets, with random interstimulus intervals between 2-5 seconds. Lapses are defined as response times greater than or equal to 355 milliseconds. The results are reported as the number of lapses with a standard deviation for the impaired condition and the non-impaired control state. More lapses suggest greater impairment.

SECONDARY OUTCOMES:
Cognition Test Battery Speed | From Study Day 2 through Study Day 6 (to include each of the three conditions: ALC, CTRL, SD1&2).
  A single variable representing response time across 10 Cognitive tasks that cover a range of cognitive domains with known cerebral representation. Subjects complete this approximately every three hours during wake. Test scores are adjusted for practice and stimulus set effects, and z-transformed based on average and standard deviation across all tests taken. Speed across cognitive domains is calculated by averaging z-scores across the 10 tests. Higher scores reflect faster speed. The final measure is reported as the least square means of the z-score.
  Scores between -0.2 and +0.2 suggest no effect on speed (0=population mean). More negative scores suggest larger negative effects (i.e. scores between -0.2 to -0.5 mean slightly slower; -0.5 to -0.8 moderately slower; scores beyond -0.8 significantly slower).
  Greater positive scores suggest larger positive effects (i.e. scores between +0.2 to +0.5 mean slightly faster; +0.5 to +0.8 moderately faster; above +0.8 significantly faster).
Cognition Test Battery Accuracy | From Study Day 2 through Study Day 6 (to include each of the three conditions: ALC, CTRL, SD1&2).
  A single variable representing accuracy across 10 Cognitive tasks that cover a range of cognitive domains with known cerebral representation. Test scores are adjusted for practice and stimulus set effects, and z-transformed based on average and standard deviation across all tests taken. Accuracy across cognitive domains is calculated by averaging z-scores across the 10 tests. Higher scores reflect better accuracy. The final measure is reported as the least square means of the z-score.
  Scores between -0.2 and +0.2 suggest no effect on accuracy (0=population mean). More negative scores suggest larger negative effects (i.e. scores between -0.2 to -0.5 mean slightly less accurate; -0.5 to -0.8 moderately less accurate; scores beyond -0.8 significantly less accurate).
  Greater positive scores suggest larger positive effects (i.e. scores between +0.2 to +0.5 mean slightly more accurate; +0.5 to +0.8 moderately more accurate; above +0.8 significantly more accurate).

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Basner, MD, PhD, MScEpi, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kiffer F, Boerma M, Allen A. Behavioral effects of space radiation: A comprehensive review of animal studies. Life Sci Space Res (Amst). 2019 May;21:1-21. doi: 10.1016/j.lssr.2019.02.004. Epub 2019 Feb 19. PMID 31101151
- [Background] Davis CM, Allen AR, Bowles DE. Consequences of space radiation on the brain and cardiovascular system. J Environ Sci Health C Toxicol Carcinog. 2021;39(2):180-218. doi: 10.1080/26896583.2021.1891825. PMID 33902387
- [Background] Basner M, Hermosillo E, Nasrini J, Saxena S, Dinges DF, Moore TM, Gur RC. Cognition test battery: Adjusting for practice and stimulus set effects for varying administration intervals in high performing individuals. J Clin Exp Neuropsychol. 2020 Jul;42(5):516-529. doi: 10.1080/13803395.2020.1773765. Epub 2020 Jun 15. PMID 32539487
- [Background] Cekanaviciute E, Rosi S, Costes SV. Central Nervous System Responses to Simulated Galactic Cosmic Rays. Int J Mol Sci. 2018 Nov 20;19(11):3669. doi: 10.3390/ijms19113669. PMID 30463349
- [Background] Basner M, Moore TM, Hermosillo E, Nasrini J, Dinges DF, Gur RC, Johannes B. Cognition Test Battery Performance Is Associated with Simulated 6df Spacecraft Docking Performance. Aerosp Med Hum Perform. 2020 Nov 1;91(11):861-867. doi: 10.3357/AMHP.5602.2020. PMID 33334406